CLINICAL TRIAL: NCT03683108
Title: Efficacy and Safety of a New Medical Device Based on Resveratrol and Carbossimetyl Beta Glucan in Treatment of Upper Airways Disease in Infancy
Brief Title: Efficacy and Safety of Resveratrol and Carbossimetyl Beta Glucan in Treatment of Upper Airways Disease in Infancy
Acronym: VIRNEO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Prof. Maria Elisabetta Baldassarre, Researcher, Policlinico Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIRNEO1
Record Dates: First submitted 2018-03-07; First posted 2018-09-25 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold | interventions — Resveratrol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol and Carbossimetyl Beta Glucan (Experimental)
  Interventions: Drug: Resveratrol and Carbossimetyl Beta Glucan
- Saline solution (Placebo Comparator)
  Interventions: Other: Saline Solution

INTERVENTIONS:
Drug: Resveratrol and Carbossimetyl Beta Glucan — Medical device based on Resveratrol and Carbossimetyl Beta Glucan. 3 drops, 4 times a day for 1 week.
  Arms: Resveratrol and Carbossimetyl Beta Glucan
Other: Saline Solution — Medical device based on Saline Solution. 3 drops, 4 times a day for 1 week.
  Arms: Saline solution

SUMMARY:
outpatient infants (0-6 months of life), affected by symptoms of upper airways disease will be randomly assigned to two type of intervention:

A: treatment group, receiving resveratrol and carbossimetyl beta glucan; B: control group, receiving saline solution.

Each subject underwent clinical history, objective examination and detection of rinovirus in the nasal secretions at enrollment, after 48 hours and after 7 and 30 days.

DETAILED DESCRIPTION:
Consecutive outpatient infants (0 - 6 months) with common cold symptoms were enrolled and randomly divided into two groups: resveratrol plus carboxymethyl-β-glucan solution or saline isotonic solution randomized treatment (3 drops in each nasal fossa, 4 time daily for seven days).

Each patient underwent clinical evaluation at enrollment, after 48 hours and after 7 and 30 days.

Common cold symptoms were specifically evaluated according to CARIFS Scale. Nasal swabs for HRV research will performed at enrollment, after 48 hours and after 7 and 30 days.

ELIGIBILITY:
Inclusion Criteria:

* common cold syndrome

Exclusion Criteria:

* main comorbidities

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Canadian Acute Respiratory Illness and Flu Scale (CARIFS) | enrollment, after 48 hours and after 7 and 30 days
  The CARIFS score consisted of 18 items each answered on a 4-point scale (no problem = 0, minor problem = 1, moderate problem = 2, major problem = 3).
  Some CARIFS items such as "headache", "sore-throat", "muscle aches or pains" were not applicable to infants. The mean of the point of all applicable items was considered as a measure of child's overall illness level.

SECONDARY OUTCOMES:
Detection of Rinovirus in the nasal secretions | after 48 hours and 7 days
  Difference in Human Rhinovirus replication will by the use of nasal swab analysis.
30-day relapses | 30-day after treatment
  Number of relapses

CONTACTS AND LOCATIONS:
Locations (1):
- Dept Of Obstetrics and Neonatology - Section of Neonatology University of Bari Policlinico Hospital, Bari, Italy

IPD SHARING:
Plan to Share IPD: No